CLINICAL TRIAL: NCT04461795
Title: A Multicenter, Open Label Study Assessing the Efficacy of AJOVY (Fremanezumab-vfrm) on Interictal Migraine Related Burden
Brief Title: Efficacy of AJOVY (Fremanezumab-vfrm) on Interictal Migraine Related Burden
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: David True (Industry)
Responsible Party: Sponsor-Investigator, David True, Medical Director, Clinvest Research, LLC
Organization: Clinvest Research, LLC (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-001TE
Record Dates: First submitted 2020-07-02; First posted 2020-07-08 (Actual); Results first posted 2022-04-13 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — erenumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- AJOVY (fremanezumab-vfrm) (Experimental): Participants received 225 mg/1.5 mL solution via single-dose prefilled syringe administered subcutaneously once every 4 weeks in the abdomen, thigh, or upper arm for 12 weeks.
  Interventions: Drug: Fremanezumab-Vfrm 225 MG/1.5 ML Subcutaneous Solution [AJOVY]

INTERVENTIONS:
Drug: Fremanezumab-Vfrm 225 MG/1.5 ML Subcutaneous Solution [AJOVY] — 225 MG/1.5 ML Subcutaneous Solution
  Other Names: fremanezumab-vfrm

SUMMARY:
This study is being conducted to evaluate the efficacy and safety of AJOVY (fremanezumab-vfrm) on interictal migraine related burden in adults.

DETAILED DESCRIPTION:
This is a single group, multicenter, open-label study with a study population of patients who meet International Classification of Headache Disorders 3rd edition (ICHD-III) criteria for migraine with or without aura and have 4 to 22 migraine days per month. This is a single-group supportive care study with one arm and no masking. A maximum of 40 participants will be enrolled to study intervention. All participants in this single-group study will complete a 4-week run-in period. After the run-in period, eligible participants will be enrolled to study intervention and enter a 12-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. willing to participate and sign informed consent;
2. ability to read and understand informed consent and study procedures, including able to use the electronic Daily Headache Diary;
3. in good general health based on investigator's judgment;
4. must be between 18 to 65 years of age, inclusive, at time of Visit 2;
5. have migraine with and/or without aura meeting the diagnostic criteria listed in the International Classification of Headache Disorders 3rd edition (ICHD-III; Appendix 5);
6. verification of headache frequency through prospectively collected baseline information during the 28-day screening/baseline phase reporting 4-22 migraine days and no more than 22 total headache days;
7. onset of migraine before age 50;
8. able to differentiate migraine from other primary headache types allowed in the study (e.g., tension-type headache);
9. stable history of migraine at least 3 months prior to screening with at least some discreet headache free periods;
10. not currently taking a migraine preventive OR has been taking a stable dose of a preventive for at least 90 days prior to screening and agrees to not start, stop, or change medication and/or dosage during the study period;

    * * participants on migraine preventive should have stable headache pattern
11. women may be included only if they have a negative pregnancy test at screening and baseline, are sterile, or postmenopausal. Women of childbearing potential (WOCBP) engaging in potentially procreative intercourse must use highly effective birth control methods for the duration of the study (i.e., starting at screening). Definitions of WOCBP, sterile and postmenopausal women, male contraception, and highly effective and acceptable birth control methods are to be determined based on investigator's judgment;
12. demonstrated compliance with the electronic Daily Headache Diary during the 28-day screening/baseline phase as defined by entry of headache data on a minimum of 23 days;
13. is willing to wear activity/sleep tracker throughout the duration of the trial;
14. has a smartphone and willing to install activity tracker app on phone.

Exclusion Criteria:

1. unable to understand the study requirements, the informed consent, or complete headache records as required per protocol;
2. pregnant, actively trying to become pregnant, or breast-feeding;
3. history of substance abuse and/or dependence that would interfere study conduction, in the opinion of the Investigator;
4. history of impaired renal function that, in the investigator's opinion, contraindicates participation in this study;
5. suffers from a serious illness, or an unstable medical condition, one that could require hospitalization, increase the risk of adverse events, or compromise data integrity (ie, likely require changes in con meds or lead to other medical investigations or treatments during the study).
6. a psychiatric condition, in the opinion of the investigator, that may affect the interpretation of efficacy and safety data or contraindicates the participant's participation in the study;
7. received nerve blocks or trigger point injections in the previous 8 weeks or plans to receive them during the study;
8. prior exposure in the last 6 months, or 5 half-lives, to biologics or drugs specifically targeting the calcitonin gene-related peptide (CGRP) pathway;
9. has failed more than 3 classes of medications for the prevention of migraine or >6 migraine preventive medications of any type due to lack of efficacy;
10. received any investigational agents within 30 days prior to Visit 1 (6 months for any investigational biological products unless previous study blind has been broken and subject was known to have received placebo);
11. plans to participate in another clinical study at any time during this study;
12. history of medication overuse of opioids or butalbital, as defined by opioid or butalbital use ≥10 days/month in each of the previous 3 months or during run-in period; Medication Overuse Headache (MOH) with other medication types will be allowed but must be documented;
13. unstable medication use for migraine prevention (changes in the last 3 months);
14. clinically relevant lab results at screening as determined by the investigator;
15. clinically relevant or significant ECG abnormalities as determined by the investigator, including ECG with QT interval corrected for heart rate (QTc) using Fridericia's correction formula (QTcF) > 500 msec;
16. history of any of the following cardiovascular conditions:

    1. Moderate to severe congestive heart failure (New York Heart Association class III or IV);
    2. Recent (within past 6 months) cerebrovascular accident, myocardial infarction, coronary stenting;
    3. Uncontrolled hypertension as defined by a confirmed systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg.
17. Subjects known to have active HIV or untreated Hepatitis C infection;
18. score of > 0 on question 9 on Patient Health Questionnaire (PHQ-9) at any visit;
19. have any other condition, that in the judgment of the investigator, would make the participant unsuitable for inclusion, or would interfere with the participant participating in or completing the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David True, Principal Investigator — Clinvest Research
Locations (2):
- United States (2):
  - StudyMetrix, City of Saint Peters, Missouri
  - Clinvest Research, LLC, Springfield, Missouri

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AJOVY (Fremanezumab-vfrm)
Started | 40
Completed | 35
Not Completed | 5
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 2
Not completed — Protocol Specified Withdrawal Criterion Met | 1

BASELINE CHARACTERISTICS:
Arm/Group | AJOVY (Fremanezumab-vfrm)
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.38 (11.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 40
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 35
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Change in Migraine Interictal Burden Scale (MIBS-4) Scores From Baseline to Weeks 4, 8, and 12.
Description: The Migraine Interictal Burden Scale (MIBS-4) is a 4-item, self-administered questionnaire which measures interictal migraine-related burden in 4 domains: impairment in work or school, impairment in family and social life, difficulty making plans or commitments, and emotional/affective and cognitive distress. Possible scores range from 0 (No interictal burden) to 12 (Severe interictal burden). Change = (Applicable Treatment Month Score - Baseline Score)
Time Frame: Baseline to Weeks 4, 8, and 12
Population: All participants enrolled and with at least one administration of investigational product (IP), will be included in this study population. The Full Analysis Population will be used to analyze the efficacy and safety endpoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- AJOVY (Fremanezumab-vfrm) - Responder: Participants received 225 mg/1.5 mL solution via single-dose prefilled syringe administered subcutaneously once every 4 weeks in the abdomen, thigh, or upper arm for 12 weeks.
  Fremanezumab-Vfrm 225 MG/1.5 ML Subcutaneous Solution [AJOVY]: 225 MG/1.5 ML Subcutaneous Solution
  Participants meeting the 50% response criteria (responders) were identified using participants' self-reported data. Responders for the purpose of this study are defined as any participant with ≥ 50% reduction in the number of migraines from baseline to at least 2 out of the 3 treatment periods.
- AJOVY (Fremanezumab-vfrm) - Non-Responder: Participants received 225 mg/1.5 mL solution via single-dose prefilled syringe administered subcutaneously once every 4 weeks in the abdomen, thigh, or upper arm for 12 weeks.
  Fremanezumab-Vfrm 225 MG/1.5 ML Subcutaneous Solution [AJOVY]: 225 MG/1.5 ML Subcutaneous Solution
  Participants not meeting the 50% response criteria (non-responders) were identified using participants' self-reported data. Non-responders for the purpose of this study are defined as any participant with < 50% reduction in the number of migraines from baseline to at least 2 out of the 3 treatment periods.
Arm/Group | AJOVY (Fremanezumab-vfrm) - Responder | AJOVY (Fremanezumab-vfrm) - Non-Responder
Number analyzed (Participants) | 21 | 19
score on a scale
  Week 4 | -1.05 (2.04) | -0.37 (1.57)
  Week 8 | -1.71 (2.59) | -0.63 (2.57)
  Week 12 | -1.71 (2.10) | -1.16 (2.81)

2. Secondary Outcome: Change in Number of Monthly Migraine Days From Baseline to Weeks 4, 8, and 12.
Description: Comparison of the mean change from baseline in the frequency of migraine headache days per 28-day period ending with the cessation of treatment month 3. A migraine headache day will be defined as a calendar day (00:00 to 23:59) with 4 or more hours of migraine headache, fulfilling International Classification of Headache Disorders-3 criteria, and/or any headache of any duration with the use of migraine-specific acute medications(s) (i.e. ergot alkaloids, ergot combinations, opioids, triptans, combination analgesics [simple analgesics combined with opioids or barbiturate with or without caffeine]). Change = (Applicable Treatment Month Score - Baseline Score)
Time Frame: Baseline to Weeks 4, 8, and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: migraine days
Arm/Group | AJOVY (Fremanezumab-vfrm) - Responder | AJOVY (Fremanezumab-vfrm) - Non-Responder
Number analyzed (Participants) | 21 | 19
migraine days
  Week 4 | -6.05 (3.41) | -0.9 (3.8)
  Week 8 | -6.71 (3.09) | -2.42 (3.34)
  Week 12 | -7.00 (3.30) | -3.53 (3.89)

3. Secondary Outcome: Change in Neuro-QoL Sleep Disturbance Short Form (SDSF) Scores From Baseline to Weeks 4, 8, and 12.
Description: The Neuro-QoL Sleep Disturbance Short Form (SDSF) is an 8-item, self-administered questionnaire which measures quality of sleep including difficulties and perception of sleep satisfaction. Possible scores range from 8 to 40, with higher scores indicating worse sleep habits. Change = (Applicable Treatment Month Score - Baseline Score)
Time Frame: Baseline to Weeks 4, 8, and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AJOVY (Fremanezumab-vfrm) - Responder | AJOVY (Fremanezumab-vfrm) - Non-Responder
Number analyzed (Participants) | 21 | 19
score on a scale
  Week 4 | -2.85 (5.20) | -4.33 (6.86)
  Week 8 | -4.30 (5.49) | -3.5 (6.87)
  Week 12 | -4.66 (5.75) | -5.23 (6.06)

4. Secondary Outcome: Change in General Self-Efficacy - Short Form (GSE-SF) Scores From Baseline to Weeks 4, 8, and 12.
Description: The General Self-Efficacy - Short Form (GSE-SF) is a 4 item, self-administered questionnaire where the participant is asked to rate their confidence in managing situations, problems, and events. Scores range from 4-20. Higher scores indicate the participant has more self-efficacy managing difficult situations. Change = (Applicable Treatment Month Score - Baseline Score)
Time Frame: Baseline to Weeks 4, 8, and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AJOVY (Fremanezumab-vfrm) - Responder | AJOVY (Fremanezumab-vfrm) - Non-Responder
Number analyzed (Participants) | 21 | 19
score on a scale
  Week 4 | -0.12 (7.02) | 2.04 (7.96)
  Week 8 | 0.46 (9.13) | 1.55 (9.00)
  Week 12 | 2.04 (7.44) | 0.98 (9.19)

5. Secondary Outcome: Change in Patient-Reported Outcomes Measurement Information System 29 (PROMIS 29) Global Pain Intensity Scores From Baseline to Weeks 4, 8, and 12.
Description: The Patient-Reported Outcomes Measurement Information System 29 (PROMIS 29) has 7 domains each with 4 questions, and then one global Pain Intensity item. The domains include: Physical Function, Anxiety, Depression, Fatigue, Sleep Disturbance, Ability to Participate in Social Roles and Activities, and Pain Interference. The global item domain is Pain Intensity. Each PROMIS domain can range from a score of 4-20, higher scores equals more of the concept being measured (e.g., more Fatigue, more Physical Function).
  The outcome measure for this endpoint is the change in the global item (Pain Intensity) from baseline. The Global Pain Intensity item can range from 0-10, with higher scores indicating more severe pain intensity. Change = (Applicable Treatment Month Score - Baseline Score)
Time Frame: Baseline to Weeks 4, 8, and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AJOVY (Fremanezumab-vfrm) - Responder | AJOVY (Fremanezumab-vfrm) - Non-Responder
Number analyzed (Participants) | 21 | 19
score on a scale
  Week 4 | -2.24 (2.63) | -0.95 (1.75)
  Week 8 | -2.29 (2.55) | -1.16 (1.77)
  Week 12 | -2.19 (2.73) | -1.74 (2.00)

6. Secondary Outcome: Change in Work Productivity and Activity Impairment - Migraine (WPAI-M) Activity Impairment Scores From Baseline to Weeks 4, 8, and 12.
Description: The Work Productivity and Activity Impairment - Migraine (WPAI-M) is a 6-item self-administered questionnaire that measures work productivity and the amount of time missed from work due to migraine. Scores are based on a percentage, so the range of scores is 0-100%, with higher scores indicating greater impairment and less productivity. Change = (Applicable Treatment Month Score - Baseline Score)
Time Frame: Baseline to Weeks 4, 8, and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AJOVY (Fremanezumab-vfrm) - Responder | AJOVY (Fremanezumab-vfrm) - Non-Responder
Number analyzed (Participants) | 21 | 19
score on a scale
  Week 4 | -20.48 (25.39) | -5.26 (23.66)
  Week 8 | -26.19 (24.59) | -7.90 (26.99)
  Week 12 | -24.76 (37.77) | -14.21 (20.90)

7. Secondary Outcome: Change in Brief Measure of Worry Severity (BMWS) Scores From Baseline to Weeks 4, 8, and 12.
Description: The Brief Measure of Worry Severity (BMWS) is a 8-item, self-administered questionnaire that measures various components of dysfunctional worry. Score range from 0-24 with higher scores indicating more worry within the participant. Change = (Applicable Treatment Month Score - Baseline Score)
Time Frame: Baseline to Weeks 4, 8, and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AJOVY (Fremanezumab-vfrm) - Responder | AJOVY (Fremanezumab-vfrm) - Non-Responder
Number analyzed (Participants) | 21 | 19
score on a scale
  Week 4 | -0.57 (2.87) | -0.05 (3.10)
  Week 8 | -0.91 (2.53) | -0.68 (4.80)
  Week 12 | -1.05 (2.33) | -1.63 (5.86)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | AJOVY (Fremanezumab-vfrm)
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 14/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AJOVY (Fremanezumab-vfrm) (N=40)
Dizziness (Nervous system disorders) | 3 (4)
Gastroenteritis (Infections and infestations) | 2 (2)
Injection site reaction (General disorders) | 5 (8)
Nausea (Gastrointestinal disorders) | 2 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to submit all manuscripts or abstracts to sponsor before submission. Sponsor will comply with the requirements for publication of study results. In accordance with standard editorial and ethical practice, the sponsor will generally support publication of multicenter studies only in their entirety and not as individual site data. In this case, a coordinating investigator will be designated by mutual agreement.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-05): https://cdn.clinicaltrials.gov/large-docs/95/NCT04461795/Prot_SAP_000.pdf